CLINICAL TRIAL: NCT07158294
Title: Digital PCR for Deep Sensitivity BCR::ABL1 Mutation Screening in CML
Brief Title: Identification of BCR::ABL1 Mutations by Digital PCR in CML
Acronym: DiP-in-CML
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CML1725
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Chronic Myeloid Leukemia (CML)
Keywords: Failure; Digital PCR; BCR:ABL1 mutation
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of BCR::ABL1 KD mutations by ddPCR in CML patients resistant to TKI (Other): Peripheral blood withdrawal for the analysis of BCR::ABL1 KD mutations by ddPCR. DdPCR results will be compared with NGS results.
  Interventions: Other: Peripheral blood withdrawal for BCR::ABL1 mutations testing

INTERVENTIONS:
Other: Peripheral blood withdrawal for BCR::ABL1 mutations testing — Peripheral blood samples taken from patients treated according to clinical practice with resistance to imatinib or 2GTKI therapy according to the ELN recommendations will be shipped to one of the reference laboratories and analyzed by ddPCR using Bio-Rad ADS assays and reagents. Samples will be analyzed in batches of suitable size. ddPCR results will be compared with NGS results. In patients positive for mutations below 20% by ddPCR (low level mutations) peripheral blood sample(s) will be collected every 3 months at subsequent follow-up visits to monitor the kinetics of mutations in relation to therapy continuation or change.

SUMMARY:
The goal of this study is to asses the ability of digital PCR (ddPCR) to detect actionable mutations in adult CML patients with failure of TKI therapy. The main objective of the study is it aims to answer is to assess whether ddPCR is at least as effective as NGS in detecting actionable (2GTKI-resistant) mutations.

To accomplish this aim, samples of participants treated according to clinical practice, will be taken and analyzed for the presence of BCR::ABL1 KD mutations by ddPCR.

DETAILED DESCRIPTION:
This is a multicenter biological study addressing the efficiency of ddPCR in detecting actionable mutations in patients with failure of TKI therapy. The study will involve 4 reference laboratories for BCR::ABL1 KD mutation testing Italian hematological centers enrolling patients and collecting samples for analysis.

Peripheral blood samples taken from patients treated according to clinical practice with resistance to imatinib or 2GTKI therapy according to the ELN recommendations will be shipped to one of the reference laboratories and analyzed by ddPCR using Bio-Rad ADS assays and reagents. Samples will be analyzed in batches of suitable size. ddPCR results will be compared with NGS results generated by reference laboratories belonging to LabNet CML network . In patients positive for mutations below 20% by ddPCR (low level mutations) peripheral blood sample(s) will be collected every 3 months at subsequent follow-up visits to monitor the kinetics of mutations in relation to therapy continuation or change.

No modification of TKI type or TKI dose will be performed on the basis of ddPCR results.

ELIGIBILITY:
Inclusion Criteria:

* molecularly confirmed diagnosis of BCR::ABL1+ CML;
* positivity for either e13a2 or e14a2 transcript;
* age ≥18 years;
* chronic phase;
* on therapy with imatinib or 2 GTKIs (dasatinib, nilotinib and bosutinib);
* candidate to TKI switch because of resistance according to the ELN recommendations OR with a confirmed warning response to 2GTKI therapy according to the ELN recommendations;
* Signed written informed consent according to ICH/EU/GCP and national local laws.

Exclusion Criteria:

* blastic phase;
* Previous allogeneic transplant or candidate to allogeneic transplant;
* on treatment with ponatinib or asciminib, investigational TKIs or non-TKI-therapy;
* switch performed or planned due to intolerance and not to resistance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Mutations detected by ddPCR | At enrollment
  The rate of actionable (2GTKI-resistant) mutations detectable by ddPCR as compared to NGS in patients with failure of TKI therapy according to the current (2020) ELN recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Simona Soverini, Principal Investigator — Department of Medical and Surgical Sciences, IRCCS Azienda Ospedaliero-Universitaria di Bologna, University of Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No